CLINICAL TRIAL: NCT05719090
Title: Acute Effects of Autoregulated and Non-autoregulated Blood Flow Restrictive Exercise on Indices of Arterial Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salisbury University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: #7
Record Dates: First submitted 2023-01-12; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Arterial Stiffness; Healthy Lifestyle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Autoregulated blood flow restriction (Active Comparator): Autoregulated BFR expands as the muscle progresses into the stretch-shortening cycle.
  Interventions: Device: Delfi Personal Tourniquet Systems
- Non-autoregulated blood flow restriction (Active Comparator): Non-autoregulated BFR does not expand as the muscle progresses into the stretch-shortening cycle.
  Interventions: Device: Delfi Personal Tourniquet Systems
- No blood flow restriction (Active Comparator): This group serves as the control group for this study
  Interventions: Device: Delfi Personal Tourniquet Systems

INTERVENTIONS:
Device: Delfi Personal Tourniquet Systems — Measure within & between differences in acute vascular compliance from pre- to post-training with autoregulated BFR, nonautoregulated BFR and no BFR conditions.

SUMMARY:
To investigate the acute effects of autoregulated (AR) and non-autoregulated (NAR) BFR exercise on indices of arterial stiffness. AR BFR training devices adjust pressure in the cuff ensuring similar pressure throughout the range of motion when the muscles are contracted (dilatated) and relaxed. NAR BFR training devices do not adjust pressure in the cuff throughout the range of motion when the muscles are contracted and relaxed which cause greater pressures at different points in the range of motion. METHODS: Following a randomized AR or NAR familiarization training session, 20 adults (23±5 years; 7 female) participated in 3 randomized treatment-order sessions with AR-BFR, NAR-BFR, and no- BFR separated by 1-week washout periods. Participants performed 4 sets of dumbbell wall squats to failure using 20% of 1 repetition maximum (1-RM) at 2-second concentric/eccentric cadence. Training limb occlusion pressure (LOP) was set at 60% of supine LOP for both the AT and NAR sessions. Testing before and immediately following the training session included ultrasonography of the carotid artery, applanation tonometry, and blood pressure acquisition. Two-way ANOVAs were used to examine the effects of treatment and the treatment-order interaction on pulse wave velocity (PWV), beta-stiffness index (β-stiff), and arterial compliance (AC). RESULTS: There were no baseline differences in CF- (carotid-femoral) PWV, CR- (carotid-radial) PWV, β-stiff, and AC (all p > 0.05). CF-PWV increased in the NAR-BFR (mean difference = 0.57±1.12 m/s, p = 0.02) and no-BFR (mean difference = 0.63±1.42 m/s, p = 0.03) groups following the exercise session. CR-PWV increased in the no-BFR (mean difference = 0.82±1.5 m/s, p = 0.03) group. And there was an interaction effect in CFPWV between AR-BFR and NAR-BFR (mean difference = 0.70±1.6 m/s, p = 0.03). CONCLUSION: These findings show acute AR-BFR training does not influence indices of arterial stiffness while acute NAR-BRF training increases central stiffness.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-40 years old
2. Physically active (> 6 months of consistent exercise training)
3. Weight stable for previous 6 months (+/-2.5 kg)
4. Female subjects only- reported regular menstrual cycles for the last 2 years

Exclusion Criteria:

1. BP>140/90 mmHg
2. BMI>40 kg/m2
3. Diabetes
4. Familial hypercholesterolemia
5. Past or current history of CHD, stroke or major CVD events. Respiratory diseases (not including asthma), endocrine or metabolic, neurological, or hematological disorders that would compromise the study or the health of the subject.
6. Women must not be pregnant, plan to become pregnant during the study, or be nursing
7. Active renal or liver disease
8. All medications and supplements that influence dependent variables
9. Recent surgery < 2 months
10. Alcohol abuse
11. Sleep apnea
12. Claustrophobia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Beta-Stiffness Index | Baseline and 10 minutes after exercise on day 1
  A measurement that compares carotid SBP and DBP with carotid systolic and diastole diameters.
Carotid-femoral pulse wave velocity | Baseline and 10 minutes after exercise on day 1
  A measurement that records the time difference between the foot of the systolic wave form as it arrives at the carotid and femoral arterial sites. It is measured with an arterial tonometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Salisbury University, Salisbury, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided